CLINICAL TRIAL: NCT07077005
Title: MavaEnEx-HOCM: Mavacamten Enables Exercise Training in Patients With Hypertrophic Obstructive CardioMyopathy. A Pilot Study
Brief Title: Mavacamten Enables Exercise in Hypertrophic Obstructive Cardiomyopathy
Acronym: MavaEnEx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, PD Dr. med. Dr. rer. nat. Simon Wernhart, Principal Investigator, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-125-S-SB
Record Dates: First submitted 2025-07-10; First posted 2025-07-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: exercise capacity; mavacamten; safety; exercise training
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to an exercise intervention group undergoing combined endurance and resistance training for 6 weeks or to a usual care group.
Who Masked: Investigator
Masking Description: The investigator will have no knowledge of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Supervised combined endurance and resistance training on top of mavacamten therapy
  Interventions: Other: Exercise training
- Usual Care (No Intervention): No supervised exercise training

INTERVENTIONS:
Other: Exercise training — Supervised, combined endurance and resistance training
  Arms: Exercise

SUMMARY:
Patients with hypertrophic obstructive cardiomyopathy and New York Heart Association Class I-II under stable treatment with mavacamten (at least 12 weeks without change of dosage) and a peak left ventricular outflow tract obstruction <50mmHg undergo either 6 weeks of structured moderate intensity endurance and resistance training (supervised, 3x/week, intervention, IT) or usual care (UC). Patients within 1 hour of travel to the training venue will be referred to IT, while those with more than 1 hour will join UC.

At baseline (visit 1, V1) and after 6 weeks of exercise intervention (visit 2, V2) all patients undergo a medical exam, resting and stress echocardiography and receive a questionnaire on the quality of life (Kansas City Cardiomyopathy Questionnaire). Cardiac biomarkers are assessed. 3 hours after stress echocardiography cardiopulmonary exercise testing is performed to measure peak oxygen consumption (VO2peak).

The primary outcome is safety. Secondary outcomes include the change of VO2peak, changes in cardiac biomarkers, resting and stress echocardiographic variables, quality of life and variables of cardiopulmonary exercise testing from V1 to V2.

DETAILED DESCRIPTION:
Patients with hypertrophic obstructive cardiomyopathy and New York Heart Association Class I-II under stable treatment with mavacamten (at least 12 weeks without change of dosage) and a peak left ventricular outflow tract obstruction <50mmHg at rest and during peak exercise undergo either 6 weeks of structured moderate intensity endurance and resistance training (supervised, 3x/week, intervention group, IT) or usual care (UC). UC will receive standard recommendations on physical activity but no supervised training. All patients receive smart watches and electrocardiograms can be triggered upon symptoms.

Patients previously treated with transcoronary septal ablation or surgical myectomy, more than low grade valve pathology during resting echocardiography, syncope or sustained ventricular tachycardia within 6 months prior to study inclusion, prior implantable cardioverter defibrillator implantation, persistent or permanent atrial fibrillation (AF) without anticoagulation for ≥4 weeks or paroxysmal or intermittent AF on screening electrocardiogram, or a corrected QT-interval (Fridericia-formula) ≥ 500 ms will be excluded. Patients with a Sudden Cardiac Death Risk Score ≥4% are excluded from the study.

Due to the rare nature of the disease and the large geographical variation, patients within 1 hour of travel to the training site will join IT, patients travelling more than 1 hour will be grouped into UC.

At baseline (visit 1, V1) and after 6 weeks of exercise intervention (visit 2, V2) all patients undergo a medical exam, resting and stress echocardiography and receive a questionnaire on the quality of life (Kansas City Cardiomyopathy Questionnaire). Cardiac biomarkers are assessed. 3 hours after stress echocardiography cardiopulmonary exercise testing (CPET) is performed to measure peak oxygen consumption (VO2peak).

The primary outcome is safety (no ventricular arrhythmias during exercise intervention or within 1 hour after completion of exercise). Secondary outcomes include changes in VO2peak, changes in cardiac biomarkers, resting and stress echocardiographic variables, quality of life and CPET variables. Physicians performing the echocardiographies and CPET analyses will be blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Diagnosis of hypertrophic obstructive cardiomyopathy
* ≥12 weeks of unchanged dosage of mavacamten
* Peak left ventricular outflow tract gradient ≤ 50 mmHg at rest and during stress echocardiography
* Left ventricular ejection fraction ≥50% at study inclusion
* New York Heart Association classes I-II

Exclusion Criteria:

* Syncope or sustained ventricular tachycardia within 6 months prior to study inclusion
* Corrected QT-interval (Fridericia-formula) ≥ 500 ms
* Paroxysmal or intermittent atrial fibrillation (AF) on screening electrocardiogram
* Persistent or permanent AF without anticoagulation for ≥4 weeks
* Previous transcoronary ablation of septal hypertrophy or surgical myectomy
* Ventricular tachycardia, significant ST-elevation or depression upon baseline cardiopulmonary exercise testing
* ≥ grade II valve insufficiencies or stenoses during resting echocardiography
* Prior implantable cardioverter defibrillator-implantation
* Sudden Cardiac Death Risk Score ≥4%

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 weeks
  Safety is defined by the abscence of adverse or serious adverse events during exercise training or within 1h of exercise termination. Adverse events include non-sustained ventricular tachycardia (nsVT) and atrial fibrillation. Serious adverse events contain hospitalization due to cardiovascular events, sustained ventricular tachycardia, nsVT with hemodynamic compromise, syncope, cardiac arrest and sudden cardiac death. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change of resting left ventricular ejection fraction | 6 weeks
  Changes of resting left ventricular ejection fraction between visit 1 and visit 2 between the exercise and usual care group.
Change of tissue Doppler velocity during peak exercise | 6 weeks
  Changes of tissue Doppler velocity (average between medial and lateral velocities) during peak exercise between visit 1 and visit 2 between the exercise and usual care group. Higher scores mean a better diastolic function.
Change of minute ventilation to carbon dioxide production | 6 weeks
  Changes of minute ventilation to carbon dioxide production between visit 1 and visit 2 between the exercise and usual care group. Higher scores mean a worse outcome.
Change of Kansas City Cardiomyopathy Score | 6 weeks
  Changes of quality of life between visit 1 and visit 2 between the exercise and usual care group. Quality of life is assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ), a difference of at least five points is considered significant. KCCQ ranges from 0 to 100 points, while 0 means worst quality of life, 100 being best quality of life.
Change of N-terminal pro-B-type natriuretic peptide and troponin I | 6 weeks
  Changes of cardiac biomarkers N-terminal pro-B-type natriuretic peptide (NTproBNP, pg/ml) and troponin I (pg/ml) between visit 1 and visit 2 between the exercise and usual care group. Higher scores mean a worse outcome.
Differences of incidence of atrial fibrillation, atrial or ventricular tachycardia on electrocardiograms | 6 weeks
  Between group differences of incidence of atrial fibrillation, atrial tachycardia or ventricular tachycardia on electrocardiograms triggered by the smart watch electrocardiograms or displayed by electrocardiograms during visits.
Change of peak oxygen consumption | 6 weeks
  Changes of peak oxygen consumption between visit 1 and visit 2 between the exercise and usual care group. A change of 1.5mL/kg/min is considered significant. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Data will be made available on reasonable request to the principal investigator

REFERENCES:
- [Result] Sachdev V, Sharma K, Keteyian SJ, Alcain CF, Desvigne-Nickens P, Fleg JL, Florea VG, Franklin BA, Guglin M, Halle M, Leifer ES, Panjrath G, Tinsley EA, Wong RP, Kitzman DW; American Heart Association Heart Failure and Transplantation Committee of the Council on Clinical Cardiology; Council on Arteriosclerosis, Thrombosis and Vascular Biology; and American College of Cardiology. Supervised Exercise Training for Chronic Heart Failure With Preserved Ejection Fraction: A Scientific Statement From the American Heart Association and American College of Cardiology. Circulation. 2023 Apr 18;147(16):e699-e715. doi: 10.1161/CIR.0000000000001122. Epub 2023 Mar 21. PMID 36943925
- [Result] Ommen SR, Ho CY, Asif IM, Balaji S, Burke MA, Day SM, Dearani JA, Epps KC, Evanovich L, Ferrari VA, Joglar JA, Khan SS, Kim JJ, Kittleson MM, Krittanawong C, Martinez MW, Mital S, Naidu SS, Saberi S, Semsarian C, Times S, Waldman CB; Peer Review Committee Members. 2024 AHA/ACC/AMSSM/HRS/PACES/SCMR Guideline for the Management of Hypertrophic Cardiomyopathy: A Report of the American Heart Association/American College of Cardiology Joint Committee on Clinical Practice Guidelines. Circulation. 2024 Jun 4;149(23):e1239-e1311. doi: 10.1161/CIR.0000000000001250. Epub 2024 May 8. Erratum In: Circulation. 2024 Aug 20;150(8):e198. doi: 10.1161/CIR.0000000000001277. PMID 38718139
- [Result] Bertero E, Canepa M, Olivotto I. Hypertrophic cardiomyopathy evolving management: American Heart Association/American College of Cardiology vs. European Society of Cardiology guidelines. Eur Heart J. 2025 Jan 21;46(4):359-361. doi: 10.1093/eurheartj/ehae507. No abstract available. PMID 39504436
- [Result] Arbelo E, Protonotarios A, Gimeno JR, Arbustini E, Barriales-Villa R, Basso C, Bezzina CR, Biagini E, Blom NA, de Boer RA, De Winter T, Elliott PM, Flather M, Garcia-Pavia P, Haugaa KH, Ingles J, Jurcut RO, Klaassen S, Limongelli G, Loeys B, Mogensen J, Olivotto I, Pantazis A, Sharma S, Van Tintelen JP, Ware JS, Kaski JP; ESC Scientific Document Group. 2023 ESC Guidelines for the management of cardiomyopathies. Eur Heart J. 2023 Oct 1;44(37):3503-3626. doi: 10.1093/eurheartj/ehad194. No abstract available. PMID 37622657
- [Result] Kim JH, Baggish AL, Levine BD, Ackerman MJ, Day SM, Dineen EH, Guseh Ii JS, La Gerche A, Lampert R, Martinez MW, Papadakis M, Phelan DM, Shafer KM; American Heart Association Leadership Committee of the Council on Clinical Cardiology; Council on Basic Cardiovascular Sciences; Council on Cardiovascular and Stroke Nursing; Council on Cardiovascular Surgery and Anesthesia; Council on Peripheral Vascular Disease; American College of Cardiology; Allen LA, Borjesson M, Braverman AC, Brothers JA, Castelletti S, Chung EH, Churchill TW, Claessen G, D'Ascenzi F, Darden D, Dean PN, Dickert NW, Drezner JA, Economy KE, Eijsvogels TMH, Emery MS, Etheridge SP, Gati S, Gray B, Halle M, Harmon KG, Hsu JJ, Kovacs RJ, Krishnan S, Link MS, Maron M, Molossi S, Pelliccia A, Salerno JC, Shah AB, Sharma S, Singh TK, Stewart KM, Thompson PD, Wasfy MM, Wilhelm M. Clinical Considerations for Competitive Sports Participation for Athletes With Cardiovascular Abnormalities: A Scientific Statement From the American Heart Association and American College of Cardiology. J Am Coll Cardiol. 2025 Mar 18;85(10):1059-1108. doi: 10.1016/j.jacc.2024.12.025. Epub 2025 Feb 20. PMID 39976316
- [Result] Basu J, Nikoletou D, Miles C, MacLachlan H, Parry-Williams G, Tilby-Jones F, Bulleros P, Fanton Z, Baker C, Purcell S, Lech C, Chapman T, Sage P, Wahid S, Sheikh N, Jayakumar S, Malhotra A, Keteepe-Arachi T, Gray B, Finocchiaro G, Carr-White G, Behr E, Tome M, O'Driscoll J, Chis Ster I, Sharma S, Papadakis M. High intensity exercise programme in patients with hypertrophic cardiomyopathy: a randomized trial. Eur Heart J. 2025 May 14;46(19):1803-1815. doi: 10.1093/eurheartj/ehae919. PMID 40037382
- [Result] Olivotto I, D'Ascenzi F. Exercise prescription in hypertrophic cardiomyopathy: Dr Lown's lesson to break taboos. Eur Heart J. 2025 May 14;46(19):1816-1818. doi: 10.1093/eurheartj/ehae659. No abstract available. PMID 40037289
- [Result] Olivotto I, Oreziak A, Barriales-Villa R, Abraham TP, Masri A, Garcia-Pavia P, Saberi S, Lakdawala NK, Wheeler MT, Owens A, Kubanek M, Wojakowski W, Jensen MK, Gimeno-Blanes J, Afshar K, Myers J, Hegde SM, Solomon SD, Sehnert AJ, Zhang D, Li W, Bhattacharya M, Edelberg JM, Waldman CB, Lester SJ, Wang A, Ho CY, Jacoby D; EXPLORER-HCM study investigators. Mavacamten for treatment of symptomatic obstructive hypertrophic cardiomyopathy (EXPLORER-HCM): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2020 Sep 12;396(10253):759-769. doi: 10.1016/S0140-6736(20)31792-X. Epub 2020 Aug 29. PMID 32871100
- [Result] Wheeler MT, Olivotto I, Elliott PM, Saberi S, Owens AT, Maurer MS, Masri A, Sehnert AJ, Edelberg JM, Chen YM, Florea V, Malhotra R, Wang A, Oreziak A, Myers J. Effects of Mavacamten on Measures of Cardiopulmonary Exercise Testing Beyond Peak Oxygen Consumption: A Secondary Analysis of the EXPLORER-HCM Randomized Trial. JAMA Cardiol. 2023 Mar 1;8(3):240-247. doi: 10.1001/jamacardio.2022.5099. PMID 36652223
- [Result] Lampert R, Ackerman MJ, Marino BS, Burg M, Ainsworth B, Salberg L, Tome Esteban MT, Ho CY, Abraham R, Balaji S, Barth C, Berul CI, Bos M, Cannom D, Choudhury L, Concannon M, Cooper R, Czosek RJ, Dubin AM, Dziura J, Eidem B, Emery MS, Estes NAM, Etheridge SP, Geske JB, Gray B, Hall K, Harmon KG, James CA, Lal AK, Law IH, Li F, Link MS, McKenna WJ, Molossi S, Olshansky B, Ommen SR, Saarel EV, Saberi S, Simone L, Tomaselli G, Ware JS, Zipes DP, Day SM; LIVE Consortium. Vigorous Exercise in Patients With Hypertrophic Cardiomyopathy. JAMA Cardiol. 2023 Jun 1;8(6):595-605. doi: 10.1001/jamacardio.2023.1042. PMID 37195701
- [Result] Maron BJ, Rowin EJ, Bonaventura J, Basso C, Corrado D, Thiene G, Churchwell AL, Basilico F, Thompson PD, Nishimura RA, Estes NAM. Commentary: Sudden death in competitive student-athletes with hypertrophic cardiomyopathy at a crossroads: Critical views on liberalizing return-to-play eligibility. Heart Rhythm. 2025 Jun 19:S1547-5271(25)02560-3. doi: 10.1016/j.hrthm.2025.06.014. Online ahead of print. No abstract available. PMID 40543859
- [Result] Pelliccia A, Sharma S, Gati S, Back M, Borjesson M, Caselli S, Collet JP, Corrado D, Drezner JA, Halle M, Hansen D, Heidbuchel H, Myers J, Niebauer J, Papadakis M, Piepoli MF, Prescott E, Roos-Hesselink JW, Graham Stuart A, Taylor RS, Thompson PD, Tiberi M, Vanhees L, Wilhelm M; ESC Scientific Document Group. 2020 ESC Guidelines on sports cardiology and exercise in patients with cardiovascular disease. Eur Heart J. 2021 Jan 1;42(1):17-96. doi: 10.1093/eurheartj/ehaa605. No abstract available. PMID 32860412